CLINICAL TRIAL: NCT02131038
Title: Non Interventional, Open Label Trial of Ectoine Containing Nasal Spray in Comparison With Cromoglycic Acid Containing Nasal Spray in Patients With Allergic Rhinitis
Brief Title: Application of Ectoine Nasal Spray in Comparison With Cromolyn Sodium Containing Nasal Spray in Patients With Allergic Rhinitis
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Rep-25
Record Dates: First submitted 2014-04-25; First posted 2014-05-06 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinitis
Keywords: Ectoine; bitop; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ectoin group: Ectoin Allergy Nasal Spray
  Interventions: Other: Medica device, drug-like
- Cromolyn group: Cromolyn sodium

INTERVENTIONS:
Other: Medica device, drug-like — Ectoin (R) Allergy Nasal Spray
  Groups: Ectoin group

SUMMARY:
This is a comparative, open label, parallel group, non interventional study to further demonstrate the effectiveness and tolerability of Ectoin Allergy Nasal Spray. In addition the effectiveness and safety shall be compared to a Cromoglycid acid containing nasal spray. The patient applies Ectoin Allergy Nasal Spray or Cromoglycid acid containing nasal spray according to the instructions for use. The observation takes place over a period of 14 days. Response to treatment is recorded at day 7 and day 14 by the physician and by the patient in a dairy at defined time intervalls.

ELIGIBILITY:
Inclusion Criteria:

* Female or male individuals ≥ 18 years
* Patients with proven Allergic Rhinitis which are treated with Ectoin Nasal Spray or -Cromoglycic acid nasal Spray during the observational period

Exclusion Criteria:

* Contra indications according to the label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in combined nasal symptom Score | Time Frame: day 1, day 7, day 14
  The change in the sum of the three different parameters nasal congestion, rhinorrhea and nasal errhine were investigated as combined score.

SECONDARY OUTCOMES:
Patient's and physician's judgment of efficacy | Day 7 and 14
  Patient and physician were asked to grade the efficacy of the treatment on a scale from 0 to 8.
Eye itching score, | Day 1, 7, 14
Epiphora score | Day1, Day 7 and Day 14
Conjunctivitis score, | Day 1, Day 7 Day 10
Palatal itching score | Day 1, Day 7, Day 14
Nasal muscle hyperplasia score | Day 1, Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Sonnemann, MD, Principal Investigator — HNO Praxis Elmshorn
Locations (1):
- HNO Praxis Elmshorn, Elmshorn, Germany